CLINICAL TRIAL: NCT05687760
Title: Effect of Bromelain Versus Calcium Hydroxide as an Intracanal Medication on the Intensity of Postoperative Pain and Bacterial Load Reduction in Necrotic Single Rooted Lower Premolars (A Randomized Clinical Trial)
Brief Title: Effect of Bromelain Versus Calcium Hydroxide as an Intracanal Medication on the Intensity of Postoperative Pain and Bacterial Load Reduction in Necrotic Single Rooted Lower Premolars
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Magy Essam Sayed El-Askary, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: magy intracanal medication
Record Dates: First submitted 2022-12-21; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Intracanal Medication; Bromelain; Calcium Hydroxide; Bacterial Load Reduction
MeSH Terms: interventions — Bromelains; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- calcium hydroxide arm (Active Comparator): intracanal medication of calcium hydroxide paste
  Interventions: Drug: Calcium hydroxide
- bromelain arm (Experimental): intracanal medication of bromelain paste (Bromelain powder with enzymatic activity of 2400 Gelatin digestion unit per Gram was mixed with saline in 1:1 proportion 1 g powder was mixed with 1 ml distilled water)
  Interventions: Biological: bromelain

INTERVENTIONS:
Biological: bromelain — is a proteolytic enzyme derived from the stem part and fruit of pineapples (Ananas comosus).used as intracanal medication
  Arms: bromelain arm
Drug: Calcium hydroxide — calcium hydroxide
  Arms: calcium hydroxide arm

SUMMARY:
the aim of the study is to compare the effect of bromelain vs calcium hydroxide as intracanal medication on intensity of pain and bacterial load in necrotic single lower premolars

DETAILED DESCRIPTION:
After diagnosing the case as pulp necrosis and confirming that the patient conforms to all eligibility criteria, the operator will enroll the patient in the study.

Treatment of all cases will be completed in two visits as follows :

1. Anesthetizing the tooth using mental nerve block technique by local anesthesia of 1.8 ml of 2% Mepivacaine HCl with 1:100,000 epinephrine (Artinibsa®; Inibsa Dental, Lliçà de Vall,Spain) .
2. Removal of Caries and/or coronal restorations completely with sterile bur and rubber dam will be applied.
3. Cleaning the operative field, including the tooth, the clamp, and rubber dam sheet, with 3% hydrogen peroxide until no further bubbling of the peroxide occurred. All surfaces will then be disinfected by a sterile cotton swab with a 5.25% sodium hypochlorite solution.
4. Preparation of access cavity using another sterile round carbide bur size 3 and Endo-z bur (Dentsply Maillefer, Ballaigues, Switzerland) .
5. After completing the access, the operative field and the pulp chamber will be cleaned and disinfected once again in the same way mentioned above. NaOCl will be then neutralized with 5% sodium thiosulfate.
6. The pre-instrumentation root canal sample (S0) will be taken as follows: a sterile paper point will be placed in the canal to soak up the fluid in the canal to a level approximately 1 mm short of the tooth apex based on diagnostic radiographs and estimated working length. The paper point will be left in the canal for at least 1 minute. Paper points will then be transferred aseptically to tubes containing sterile brain heart infusion (BHI) broth.
7. Confirming the patency of the root canals using stainless steel hand K-files size #10 and #15(K-Files, MANI, INC., Industrial Park, Utsunomiya, Tochigi, Japan) Working length will be determined using an electronic apex locator(Root ZX, J. Morita USA, Irvine, CA) then confirmed radiographically to be 1 mm shorter than radiographic apex.
8. Mechanical preparation will be done using M PRO rotary files in an endodontic motor (X-Smart, Dentsply Maillefer, USA) The first file (18/.09) will be used as an orifice opener for two thirds of the working length followed by (20/.04) and (25/.06) for the full working length and finally (35/.04). In-and-out motions will be applied with stroke lengths not exceeding 3 mm in the cervical, middle, and apical thirds until attaining the established WL. The first file is used with a continuous rotary motion at a speed of 500rpm and torque of 3Ncm. The second, third and fourth files are used with a speed of 300 rpm and torque of 1.5Ncm. The canal will be irrigated and recapitulated after the use of each instrument.
9. The canal will be thoroughly irrigated with 2.5% sodium hypochlorite root canal irrigant (5ml for 1 min) using disposable plastic syringe with side vented needle gauge 30 (Steri irrigation tips; Diadent, Chungcheongbuk-do, Korea) reaching 1 mm short of the working length. All teeth will receive the same volume of irrigant (5 ml prior to instrumentation, 5 ml between each file and 5 ml as final flush after root canal instrumentation to reach a total volume of 25 ml in total).
10. Post-instrumentation sample (S1) will be taken as previously mentioned.
11. The patients will then be assigned into two groups :

    In the intervention groups, Bromelain paste (Bromelain powder with enzymatic activity of 2400 Gelatin digestion unit per Gram was mixed with saline in 1:1 proportion 1 g powder was mixed with 1 ml distilled water) will be placed inside the canals using sterile plastic syringe with needle gauge 27 without binding 1mm shorter than working length . The access cavities were closed using sterile cotton pellet and intermediate restorative material .

    In the control group, Ca(OH)29will be placed inside the canals using sterile plastic syringe with needle gauge 27 without binding 1 mm shorter than working length .The access cavities were closed using sterile cotton pellet and intermediate restorative material .
12. Patients will be asked to record their pain level after the first visit on Numeric Rating Scale (NRS) at 6, 12, 24, 48 hours.(Appendix V)
13. Each patient will be given a chart to record postoperative swelling. If swelling was recorded, the patient will be appointed for clinical examination to assess the severity by blinded assessor in a swelling rating scale and to determine if systemic antibiotics (Augmentin 625mg/8 hours/5 days) or drainage would have been needed.
14. In the recall appointment after 1 week. Rubber dam will be applied then intracanal medication will be removed using copious irrigation and fanta AF max rotary file (#25 0.04) and tooth will be disinfected as before. The previously sampled canal will be re-entered, flushed with copious saline irrigation and a third sample (S-2) will be taken. After the sampling, final flush with 2.5% NaOCL and 17% EDTA will be done in both groups. Master cones of (0.40) taper gutta-percha(Meta Biomed Co., Ltd, Korea) will be fitted to the working length and a radiograph will be taken to ensure proper length. Obturation will be done by modified single cone technique using epoxy resin sealer(Adseal, Meta Biomed CO.,LTD, Korea)and 4% taper gutta percha cones together with auxillary cones.
15. The tooth will be sealed by temporary restoration ,Then the details of the endodontic procedure for each patient will be recorded in the patient's procedure chart (Appendix IV) .
16. The patient will be instructed to return to complete the treatment procedures until placing a full-coverage restoration.
17. In case of severe pain or persisting pain patients are instructed to take prescribed analgesic (Ibuprofen 400mg), not to take it less than 6 hours apart

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are free from any physical or mental handicapping condition with no underlying systemic disease (ASA I or II) .
2. Age between 25-50 years old.
3. Males & Females.
4. Patients who can understand pain scale and can sign the informed consent.
5. Mandibular Single rooted premolars, having single root canal:

   * Diagnosed clinically with pulp necrosis.
   * Absence of spontaneous pulpal pain.
   * Positive pain on percussion denoting apical periodontitis.
   * Slight widening in the periodontal membrane space with or without periapical radiolucency radiographically.
   * Normal occlusal contact with opposing teeth

Exclusion Criteria:

* Medically compromised patients: Pain levels and healing following treatment would be compromised as these patients have shown higher incidence of pain and lower healing rate.
* Pregnant women: Avoid radiation exposure, anesthesia, and medication.
* If antibiotics have been administrated by the patient during the past 12 hours preoperatively might alter their pain perception.
* Patients reporting bruxism or clenching: Avoid further pressure on an already inflamed tooth inducing subsequent irritation and inflammation.
* Teeth that shows association with acute periapical abscess and swelling: Need special treatment steps which could involve additional visits with incision and drainage. Also, it could influence initiation and progression of postoperative pain.
* Greater than grade I mobility or pocket depth greater than 5mm. Need special surgical and/or periodontal therapy.
* No restorability: Hopeless tooth.
* Immature teeth.
* Radiographic evidence of external or internal root resorption.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-10 (Estimated); Primary Completion 2023-02-10 (Estimated); Study Completion 2023-02-10 (Estimated)

PRIMARY OUTCOMES:
postoperative pain intensity | 6 hours post-instrumentation
  measured using Numerical rating scale
postoperative pain intensity | 12 hours post-instrumentation
  measured using numerical rating scale
postoperative pain intensity | 24 hours post-instrumentation
  measured using numerical rating scale
postoperative pain intensity | 48 hours post-instrumentation
  measured using numerical rating scale

SECONDARY OUTCOMES:
bacterial load reduction | immediately after access preparation and pre- instrumentation.
  using Colony forming unit (CFU )
enterococcal bacterial count | immediately after access preparation and pre- instrumentation.
  using Colony forming unit (CFU )
bacterial load reduction | immediately after instrumentation
  using Colony forming unit (CFU )
enterococcal bacterial count | immediately after instrumentation
  using Colony forming unit (CFU )
bacterial load reduction | 1 week after intracanal medicament placement
  using Colony forming unit (CFU )
enterococcal bacterial count | 1 week after intracanal medicament placement
  using Colony forming unit (CFU )
Incidence of inter- appointment swelling | Up to 48 hours post- operatively
  using binary chart (yes or no)

IPD SHARING:
Plan to Share IPD: Undecided